CLINICAL TRIAL: NCT05545358
Title: Experimental Study of the Neural Bases of Phantom Pain After Amputation and Their Modification by Proprioceptive Training: MRI Study of the Brain and Spinal Cord
Brief Title: Neural Bases of Phantom Pain After Amputation
Acronym: Phantom limb
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PPRC09; 2021-A01733-38 (Other: IDRCB)
Record Dates: First submitted 2022-09-12; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Phantom Pain
Keywords: fMRI; spinal fMRI
MeSH Terms: conditions — Phantom Limb | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Amputees with phantom pain: Adult patients who have been amputated for more than 2 years and have chronic phantom pain
  Interventions: Other: Questionnaires; Device: Brain and Spinal Cord functional Magnetic Resonance Imaging; Other: Proprioceptive training
- Amputees without phantom pain: Adult patients who have been amputated for more than 2 years and do not have chronic phantom pain
  Interventions: Other: Questionnaires; Device: Brain and Spinal Cord functional Magnetic Resonance Imaging
- Healthy participants: Healthy adult participants with no neurological history
  Interventions: Device: Brain and Spinal Cord functional Magnetic Resonance Imaging; Other: Proprioceptive training

INTERVENTIONS:
Other: Questionnaires — Short-Form McGill Pain Questionnaire (SF-MPQ) Pain Disability Index (PDI) Prosthesis Evaluation Questionnaire (PEQ) Psychological Inflexibility to Pain Scale (PIPS) Chronic Pain Acceptance Questionnaire (CPAQ) Cognitive Difficulties Scale (CDS) Amputee Body Image Scale (ABIS) Trinity Amputation and Prosthesis Experience Scales (TAPES) Pain Catastrophizing Scale (PCS) Hospital Anxiety and Depression Scale (HAD) Credibility/Expectancy Questionnaire (CEQ) Short-Form Edinburgh Handedness Inventory (SF-EHI) Patient's Global Impression of Change (PGIC)
  Groups: Amputees with phantom pain; Amputees without phantom pain
Device: Brain and Spinal Cord functional Magnetic Resonance Imaging — Brain and Spinal Cord functional Magnetic Resonance Imaging
Other: Proprioceptive training — Proprioceptive muscular training via a mechanical vibration of low amplitude and frequency between 60 and 80 Hz applied to the tendons.
  Groups: Amputees with phantom pain; Healthy participants

SUMMARY:
The amputation of a limb results in chronic pain associated with the lost limb in the majority of patients, which persists over time. Despite a large number of studies conducted in an attempt to elucidate the neural basis of phantom pain, these are still not elucidated and current treatments often fail to relieve patients' pain.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years old
* For the "amputees with phantom pain" group: patients who have been amputated for more than 2 years and have chronic phantom pain
* For the "amputees without phantom pain" group: patients who have been amputated for more than 2 years and do not have chronic phantom pain
* For the "healthy participants" group: healthy participants with no neurological history

Exclusion Criteria:

* Clinically significant pathology (gastrointestinal, renal, hepatic, endocrine, cardiovascular or respiratory)
* Progressive psychiatric or neurological pathology
* On psychotropic medication
* Pregnant or nursing woman
* Inadequate level of French language

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is composed of :
  * patients who have been amputated for more than 2 years and have chronic phantom pain;
  * patients who have been amputated for more than 2 years and do not have chronic phantom pain;
  * healthy participants with no neurological history. The patients will be recruited from the cohort of amputee patients followed by the Physical Medicine and Rehabilitation departments of the Hôpital d'Instruction des Armées Laveran, the Hôpital d'Instruction des Armées Desgenettes and the CHU de Saint-Etienne.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in brain activity, measured through fMRI, following proprioceptive training | Up to 3 months
  Brain activity (BOLD hemodynamic response) will be measured via fMRI before and after proprioceptive training sessions.
Change in spinal cord activity, measured through spinal fMRI, following proprioceptive training | Up to 3 months
  Spinal cord activity (BOLD hemodynamic response) will be measured via spinal fMRI before and after proprioceptive training sessions.